CLINICAL TRIAL: NCT02455765
Title: Glycemic Response of Co-ingesting Carbohydrate and Amino Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: Cerebos Asia Pacific Pte Ltd (Unknown)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2014/00366
Record Dates: First submitted 2015-05-21; First posted 2015-05-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Metabolic Diseases
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- White rice control (Experimental): Subjects will consume white rice as control (50g carbohydrate)
  Interventions: Other: Rice and Amino Acid mixtures
- co-ingest low dose of amino acid (Experimental): Subjects will receive 68 ml of amino acid mixture together with white rice
  Interventions: Other: Rice and Amino Acid mixtures
- co-ingest high dose of amino acid (Experimental): Subjects will receive 136 ml of amino acid mixture together with white rice
  Interventions: Other: Rice and Amino Acid mixtures
- pre-load low dose15 min (Experimental): Subjects will receive 68 ml of amino acid mixture 15 min before consumption of white rice
  Interventions: Other: Rice and Amino Acid mixtures
- pre-load low dose 30 min (Experimental): Subjects will receive 68 ml of amino acid mixture 30 min before consumption of white rice
  Interventions: Other: Rice and Amino Acid mixtures
- pre-load high dose 15 min (Experimental): Subjects will receive 136 ml of amino acid mixture 15 min before consumption of white rice
  Interventions: Other: Rice and Amino Acid mixtures
- pre-load high dose 30 min (Experimental): Subjects will receive 136 ml of amino acid mixture 30 min before consumption of white rice
  Interventions: Other: Rice and Amino Acid mixtures

INTERVENTIONS:
Other: Rice and Amino Acid mixtures — Rice and amino acid mixture

SUMMARY:
The study will investigate if consumption of amino acid mixtures results a change in glycemic response of carbohydrate (white rice) and insulinemic response at different doses and timing (before consumption of carbohydrate).

DETAILED DESCRIPTION:
Healthy male subjects will be served with amino acid mixtures in combinations of two doses and three time points along with white rice as control. The combinations were either low or high levels of amino acid mixtures. This was consumed together or 15 min, 30 min before consumption of white rice. Postprandial blood glucose and plasma insulin concentrations were measured at fasting and every 15 min after consumption of treatment meal until 60 min after the consumption of white rice. Subsequent blood sample were taken at 30 min interval until 210min. The glucose and insulin in the blood will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Chinese ethnicity
* Age between 21-50 years
* Body mass index (BMI) between 18-24.9 kg/m2
* Waist circumference ≤ 90 cm for men
* Normal blood pressure (<120/80 mmHg)
* Fasting blood glucose < 6 mmol/L

Exclusion Criteria:

* dislike the consumption of Essence of Chicken
* participating in competitive sports
* allergic to amino acids and rice
* metabolic diseases (such as diabetes, hypertension and the metabolic syndromes)
* Glucose-6-Phosphate-Dehydrogenase (G6PD) Deficiency
* on prescription medication
* smokers

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2014-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Glycemic response | 210 minutes post consumption of carbohydrate
  Blood glucose will be assessed via finger prick during fasting and every 15 minutes for the first 60 min after the consumption white rice and subsequently every 30 min interval until 210 min
Insulinemic response | 210 minutes post consumption of carbohydrate
  Plasma insulin will be assessed via finger prick during fasting and every 15 minutes for the first 60 min after the consumption white rice and subsequently every 30 min interval until 210 min